CLINICAL TRIAL: NCT00384228
Title: A Phase I/II Multicenter, Dose-escalation Study of Oral Nilotinib on a Continuous Daily Dosing Schedule in Adult Patients With Imatinib-resistant or Imatinib-intolerant CML, or Relapse/Refractory Ph+ALL
Brief Title: A Phase l/ll Study of AMN107 in Adult Patients With Glivec-intolerant CML or Relapsed-refractory Ph+ALL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107A1101
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2012-04

CONDITIONS: Chronic Myelogenous Leukemia; Acute Lymphoblastic Leukemia (Philadelphia Chromosome Positive)
Keywords: Chronic Myelogenous Leukemia; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — nilotinib

ARMS (1):
- Nilotinib (Experimental)
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib
  Other Names: AMN107

SUMMARY:
This study will investigate if nilotinib provides an improved safety and efficacy profile over that seen in patients receiving Imatinib.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as Ph+ ALL who are either relapsed after or refractory to standard therapy
* Diagnosed as CML in blast crisis or accelerated phase or chronic phase who are resistant or intolerant to imatinib
* Performance status is normal or ambulatory and capable of all self-care Exclusion Criteria
* A history of significant or serious uncontrolled cardiovascular disease
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of nilotinib
* Patients who are pregnant or breast feeding, or adults of reproductive potential not employing an effective method of birth control

Exclusion Criteria:

* Cytopathologically confirmed CNS infiltration NB: in absence of suspicion of CNS involvement, lumbar puncture is not required
* Impaired cardiac function, including any one of the following

  * LVEF < 45% as determined by echocardiogram
  * Complete left bundle branch block
  * Use of a cardiac pacemaker
  * ST depression of > 1mm in 2 or more leads and/or T-wave inversions in 2 or more contiguous leads
  * Congenital long QT syndrome
  * History of or presence of significant ventricular or atrial tachyarrhythmias
  * Clinically significant resting bradycardia (< 50 beats per minute)
  * QTc > 480 msec on screening ECG (using the QTcF formula)
  * Right bundle branch block plus left anterior hemiblock, bifascicular block
  * Myocardial infarction within 3 months prior to starting AMN107
  * Uncontrolled angina pectoris
* Other clinically significant heart disease (e.g., congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of AMN107 (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Use of therapeutic warfarin
* Acute or chronic liver or renal disease considered unrelated to tumor (e.g., hepatitis, cirrhosis, renal insufficiency, etc.)
* Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes, active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
* Treatment with any hematopoietic colony-stimulating growth factors (e.g., G-CSF) ≤ 1 week prior to starting study drug.
* Patients who are currently receiving treatment with any of the medications listed in (cf. Post-text suppl. 5) that cannot be either discontinued or switched to a different medication prior to starting study drug. The medications listed in (cf. Post-text suppl. 5) have the potential to prolong the Q-T interval.
* Patients who have received chemotherapy ≤ 1 week or who are within 5 half-lives of their last dose chemotherapy (6 weeks for nitrosurea or mitomycin-C) prior to starting study drug or who have not recovered from side effects of such therapy. Hydroxyurea is permitted at the investigator's discretion prior to enrollment.
* Patients who have received Glivec® ≤ 1 week or who have not recovered from side effects of such therapy.
* Patients who have received immunotherapy ≤ 1 week prior to starting study drug or who have not recovered from side effects of such therapy.
* Patients who have received any investigational drug (excluding STI571/Glivec) ≤ 4 weeks or investigational cytotoxic agent within 1 week (or who are within 5 half-lives of a previous investigational cytotoxic agent) prior to starting study drug or who have not recovered from side effects of such therapy.
* Patients who have received wide field radiotherapy ≤ 4 week or limited field radiation for palliation ≤ 2 week prior to starting study drug or who have not recovered from side effects of such therapy.
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Patients who are pregnant or breast feeding, or adults of reproductive potential not employing an effective method of birth control. (Women of childbearing potential must have a negative serum pregnancy test within 48 hrs prior to administration of AMN107). Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug
* Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory)
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention.
* Patients unwilling or unable to comply with the protocol

Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-05; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Safety evaluation assessed by dose limiting toxicity within first cycle of 28 day treatment and AEs within 3 cycles | every first 28 days
Pharmacokinetic (PK) profile of single and multiple doses | day 1 and 15 of cycle 1,day 6, 8, 10, 12, 22 and 28 of cycle 1, day 15 of cycle 2

SECONDARY OUTCOMES:
Anti-leukemic activity within 3 cycles of 28 days treatment | Day 28 cycle 1, 2 and 3, at the time of disease progression, and at the time of study completion
Bone marrow and/or blood assessments to detect the presence of Bcr-Abl transcript and mutational analysis of Bcr-Abl before, during and after therapy. | Day 28 cycle 1, 2 and 3, at the time of disease progression, and at the time of study comp

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Tokyo, Japan

REFERENCES:
- [Derived] Lange T, Ernst T, Gruber FX, Maier J, Cross M, Muller MC, Niederwieser D, Hochhaus A, Pfirrmann M. The quantitative level of T315I mutated BCR-ABL predicts for major molecular response to second-line nilotinib or dasatinib treatment in patients with chronic myeloid leukemia. Haematologica. 2013 May;98(5):714-7. doi: 10.3324/haematol.2012.068890. Epub 2012 Oct 12. PMID 23065514
- [Derived] le Coutre P, Ottmann OG, Giles F, Kim DW, Cortes J, Gattermann N, Apperley JF, Larson RA, Abruzzese E, O'Brien SG, Kuliczkowski K, Hochhaus A, Mahon FX, Saglio G, Gobbi M, Kwong YL, Baccarani M, Hughes T, Martinelli G, Radich JP, Zheng M, Shou Y, Kantarjian H. Nilotinib (formerly AMN107), a highly selective BCR-ABL tyrosine kinase inhibitor, is active in patients with imatinib-resistant or -intolerant accelerated-phase chronic myelogenous leukemia. Blood. 2008 Feb 15;111(4):1834-9. doi: 10.1182/blood-2007-04-083196. Epub 2007 Nov 29. PMID 18048643
- See also: Results for CAMN107A1101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2952